CLINICAL TRIAL: NCT05097898
Title: Évaluation de la Congestion en Ambulatoire Chez Les Patients Atteints d'Insuffisance Cardiaque Chronique à Fraction d'éjection préservée. CHF-COV Preserved (Chronic Heart Failure With Preserved Ejection Fraction - COngestion eValuation)
Brief Title: Chronic Heart Failure With Preserved Ejection Fraction - COngestion eValuation
Acronym: CHF-COV-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr. Nicolas GIRERD, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020PI145-3
Record Dates: First submitted 2021-10-11; First posted 2021-10-28 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-03

CONDITIONS: Chronic Heart Failure; Preserved Ejection Fraction
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with chronic HFpEF coming for scheduled day hospitalization or consultation (Experimental): * Clinical examination focusing on congestion
  * Cardiac, pulmonary, peritoneal, jugular and renal venous Doppler ultrasounds
  * Blood sample retrieved for biological assessment and biobanking
  * Telephone follow-up
  Interventions: Procedure: Clinical examination centered on congestion; Procedure: Cardiac, pulmonary, peritoneal, jugular and renal Doppler ultrasounds and liver elastography; Procedure: Blood and urine sample retrieved for biological assessment and biobanking; Other: Telephone follow-up; Behavioral: Kansas City Cardiomyopathy Questionnaire (KCCQ)

INTERVENTIONS:
Procedure: Clinical examination centered on congestion — Clinical examination centered on congestion (including the EVEREST, Ambrosy and ASCEND score) will be performed during day hospitalization or consultation
Procedure: Cardiac, pulmonary, peritoneal, jugular and renal Doppler ultrasounds and liver elastography — Cardiac, vena cava, pulmonary, peritoneal, jugular and renal Doppler ultrasounds and liver elastography will be performed during day hospitalization or consultation/ peritoneal, jugular and renal Doppler ultrasounds and liver elastography are optional/Cardiac echo is optional for patients included in consultation
Procedure: Blood and urine sample retrieved for biological assessment and biobanking — Blood sample retrieved for biological assessment and biobanking will be performed during day hospitalization or consultation/ Urine analysis is optional for patients included in consultation
Other: Telephone follow-up — Telephone follow-up will be performed 3, 12 and 24
Behavioral: Kansas City Cardiomyopathy Questionnaire (KCCQ) — Questionnaire centered on patient's quality of life at discharge and 3, 12 and 24 months after discharge

SUMMARY:
Heart failure (HF) is a significant cause of death and the leading cause of hospitalization in patients over 65 years of age. Congestion is the main source of symptoms and the leading cause of hospitalization for HF. Furthermore, congestive signs identified in asymptomatic patients are associated with the risk of developing symptomatic HF. The literature supports a multi-modality / integrative evaluation of congestion, combining clinical examination, laboratory results and ultrasound evaluation.

The main objective of the CHF-COV Preserved study is to identify congestion markers (clinical, biological and ultrasound) quantified during a consultation or day hospitalization for the monitoring of chronic HF with preserved left ventricular ejection fraction that are associated with the risk of all-cause death, hospitalization for acute HF or IV diuretics injection in a day hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic acute heart failure with preserved ejection fraction admitted in hospital for scheduled day hospitalization or consultation
* Patient with preserved left ventricular ejection fraction (≥50%).
* Age ≥18 years
* Patients having received complete information regarding the study design and having signed their informed consent form.
* Patient affiliated to or beneficiary of a social security scheme

Exclusion Criteria:

* Comorbidity for which the life expectancy is ≤ 3 months
* Dialysis patient (peritoneal dialysis or hemodialysis) or patients with glomerular filtration rate <15 ml/min/m2 at inclusion.
* History of lobectomy or pneumonectomy lung surgery
* Severe pulmonary or pleural pathology preventing reliable acquisition of lung ultrasound images: severe emphysema, chronic pleurisy, pulmonary fibrosis, etc.
* Pregnant woman, parturient or nursing mother
* Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
* Adult person who is unable to give consent
* Person deprived of liberty by a judicial or administrative decision,
* Person subject to psychiatric care pursuant to Articles L. 3212-1 and L. 3213-1 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2028-12-10 (Estimated); Study Completion 2029-06-10 (Estimated)

PRIMARY OUTCOMES:
Rate of death from all causes | 24 months after inclusion
  composite endpoint : rate of death from all causes, hospitalisation for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following inclusion (with outcome 2 and 3)
Rate of hospitalisation for acute heart failure | 24 months after inclusion
  composite endpoint : rate of death from all causes, hospitalisation for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following inclusion (with outcome 1 and 3)
Rate of day-hospital or in-home IV diuretics injection for acute HF | 24 months after inclusion
  composite endpoint : rate of death from all causes, hospitalisation for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following inclusion (with outcome 1 and 2)

SECONDARY OUTCOMES:
Number of B-lines measured in lung echography | At baseline
Rate of death from all causes | 24 months after inclusion
  composite endpoint : Rate of death from all causes or hospitalisation for acute heart failure 24 months after inclusion (with outcome 6)
Rate of hospitalisation for acute heart failure | 24 months after inclusion
  composite endpoint : Rate of death from all causes or hospitalisation for acute heart failure 24 months after inclusion (with outcome 5)
Rate of death from all causes | 24 months after inclusion
Rate of hospitalisation for acute heart failure | 24 months after day hospitalization
  composite endpoint: Rate of hospitalisation for acute heart failure or day-hospital/in-home IV diuretics injection for acute HF 24 months after inclusion (with outcome 9)
Rate of day-hospital or in-home IV diuretics injection for acute HF | 24 months after inclusion
  composite endpoint: Rate of hospitalisation for acute heart failure or day-hospital/in-home IV diuretics injection for acute HF 24 months after inclusion (with outcome 8)
Rate of hospitalisation for cardiovascular reason | 24 months after inclusion
Rate of death from all causes | 24 months after inclusion
  composite endpoint : Rate of death from all causes or hospitalisation for acute heart failure 24 months after inclusion (with outcome 12)
Rate of hospitalisation for acute heart failure | 24 months after inclusion
  composite endpoint : Rate of death from all causes or hospitalisation for acute heart failure 24 months after inclusion (with outcome 11)
Rate of cardiovascular death | 24 months after inclusion
NYHA (New York Heart Association) class measured | 3, 12 and 24 months after inclusion
Natriuretic peptides | At baseline
  BNP or Nt-Pro BNP
Renal function | At baseline
  Assessed by glomerular filtration rate
Plasma volume | At baseline
  Calculated from haemoglobin and haematocrit value
Rate of bilirubin | At baseline
Rate of ASAT | At baseline
Rate of ALAT | At baseline
Rate of V factor | At baseline
Blood potassium concentration | At baseline
Liver elastography value | At inclusion
  Measured with Fibroscan®
Quality of life assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) | At inclusion and 3, 6 and 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No